CLINICAL TRIAL: NCT03881579
Title: Supportive Care for Cognitively Impaired Patients and Families
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, VJ Periyakoil, Director. Palliative Care Education & Training, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 48000; R01AG062239-01 (NIH)
Record Dates: First submitted 2018-10-08; First posted 2019-03-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Dementia; Primary Palliative Care; Mild Cognitive Impairment
Keywords: palliative; supportive; MCI; palliative care; supportive care; serious illness; RCT; randomized clinical trial; mild cognitive impairment; primary palliative care
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: patients will be randomized to one of two groups:
  1. (usual care) or (2). enhanced usual care i.e. usual care plus supportive care provided by a trained and supervised nurse
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed by blinded research associates
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Other): one random half of patients will receive usual care
  Interventions: Behavioral: nurse-led supportive care assessment
- intervention arm (Experimental): one random half of patients will receive enhanced usual care (usual care plus nurse-led supportive care intervention)
  Interventions: Behavioral: nurse-led supportive care assessment

INTERVENTIONS:
Behavioral: nurse-led supportive care assessment — Trained project nurses will conduct systematic assessment and provide coaching to patients in the experimental arm

SUMMARY:
Currently almost 5 million Americans suffer from the distressing symptoms related to dementia and this number that will triple by 2050. The overall goals of the proposed project are to evaluate, in community dwelling Alzheimer's Disease Research Center participants the benefits of a 12-month nurse-led early palliative intervention on symptoms, quality of life, health care resource use. The relevance of this research to public health is that there is an urgent need to improve the palliative care of persons with dementia living in the community. This study will contribute substantially to that effort.

DETAILED DESCRIPTION:
200 persons who participate in the Stanford ADRC will be recruited and randomized 100 each to usual care (UC) or {usual care plus an early palliative care intervention} (EPC) to be delivered by a nurse over a twelve-month period. The EPC will include one nurse-led palliative consult for a two-hour virtual session followed by 11 monthly 30-minute phone/video sessions plus usual care. The study aims are to determine whether EPC will lead to (a) eliciting and alleviating the supportive care needs of patients, (b) elicit their goals of care and help them complete and sign (with witnesses) their Advance Directives and the POLST (signed by the patient/proxy and their doctor) upload these into the electronic health records. Exploratory outcomes will include health resource use (e.g. hospital admissions and days, emergency visits) for the participants and caregiver burden for their caregivers. Mixed-methods framework will be utilized to analyze the audiotapes of the encounters between the research nurse and the patient during the twelve intervention sessions and to assess whether the information that is provided to participants differs by patient ethnicity and cognitive levels.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in the Stanford Alzheimers Disease Research Center (SADRC).
* All caregivers enrolled in the Stanford Alzheimers Disease Research Center (SADRC).

Exclusion Criteria:

1. Institutionalized (not a community dweller) at the time of entry into the study;
2. Have severe dementia and are incapable of responding to the outcome measures at baseline. 3. Participants who live alone and don't have a proxy will be excluded only if they are deemed as lacking the capacity to provide informed consent at the time of entry into the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify the number of participants who express supportive care needs in both arms. | Day 0, 4 months, one year
  Only the participants randomized to the intervention arm will receive the nurse-led supportive care intervention (one session per month over a twelve-month period).
  We hypothesize that compared to the control arm, many more patients in the intervention arm will express supportive needs and have them fulfilled by the study nurses.
Change in Zarit Caregiver Burden scores over time: | Day 0, 4 months, one year, 18 months
  The Zarit Burden Interview contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always) . The factor structure is a two-factor model, addressing personal strain and role strain. The investigators will assess change in Zarit scores between three points in time : on study entry, one year later and two year later.
Completion of goals of care discussion and documentation of advance directives (AD) and the Physicians Orders for Life Sustaining Treatment (POLST) in the electronic health records. | Day 0, 4 months, one year, 18 months
  In both arms the investigators will track the completion, signage and documentation of advance directives and the POLST. We will monitor the EHR to track if the doctor documents goals of care in the chart.AD has to be signed by the patient or proxy and witnessed by two qualifying witnesses. The POLST has to be signed by the patient/proxy and the doctor. Both forms have to be uploaded into the electronic health records.

SECONDARY OUTCOMES:
Differences in Edmonton Symptoms Assessment Scale (ESAS) scores | Day 0, 4 months, one year, 18 months
  The ESAS is designed to assist in the assessment of nine symptoms common in patients: pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, wellbeing and shortness of breath, (there is also a line labelled "Other Problem"). The severity at the time of assessment of each symptom is rated from 0 to 10 on a numerical scale, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity. The investigators will assess change in ESAS score of all participants at baseline, months 4, 12 and 18. The investigators hypothesize that patients with cognitive impairment will have higher scores than those with normal cognition. The investigators will also determine changes in the ESAS score (if any) over time.
Change in Patient Activation Measure over time | one year, two years
  3-item survey that assesses a person's underlying knowledge, skills and confidence integral to managing his or her own health and healthcare.
  PAM segments individuals into one of four activation levels along an empirically derived 100-point scale. Each level provides insight into an extensive array of health-related characteristics, including attitudes, motivators, and behaviors. Individuals in the lowest activation level do not yet understand the importance of their role in managing their own health, and have significant knowledge gaps and limited self-management skills. Individuals in the highest activation level are proactive with their health, have developed strong self-management skills, and are resilient in times of stress or change. PAM measures patient activation and agency: The investigators will assess changes in activation scores in ESAS scores between three points in time : on study entry, one year later and two year later.

CONTACTS AND LOCATIONS:
Overall Officials: VJ Periyakoil, MD, Principal Investigator — Stanford University
Locations (1):
- VJ Periyakoil, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
this will depend on if patients consent or not for release of data
Supporting Information: Study Protocol, SAP
Time Frame: after study completion
Access Criteria: by emailing study team